CLINICAL TRIAL: NCT05264285
Title: Exploring the Relationship Between Mitochondrial Health and Hemodynamic Instability Related to Renal Replacement Therapy in Critically Ill Patients
Brief Title: Mitochondrial Health and Hemodynamic Instability Related to Renal Replacement Therapy in Critically Ill Patients
Acronym: MitoHIRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Edward Clark, Clinical investigator, Ottawa Hospital Research Institute
Other Study IDs: 20200699-01H
Record Dates: First submitted 2021-11-23; First posted 2022-03-03 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Acute Kidney Injury (AKI)
Keywords: Renal replacement therapy (RRT); Slow low-efficiency dialysis (SLED); Metabolites; Nicotinamide adenine dinucleotide (NAD+); Hemodynamic instability related to RRT (HIRRT); Intensive care unit (ICU)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological specimen collection of pre-and post-dialysis blood samples for up to 5 consecutive SLED treatments. Dialysate samples will be collected from the first 30 patients' initial SLED treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal replacement therapy is a life-saving treatment for patients who have sudden and severe kidney failure. However, some of these patients blood pressure who receive this treatment could become unstable, thus resulting in more injuries to their kidneys and may limit the ability of kidney recovery. In order to mitigate the instability in blood pressure, the mitochondrial functions should be studied. Mitochondria are organelles within our bodies' cells that serve as the main source of energy for cell function. Kidney cells have many of these organelles and when they are damaged, it could contribute to kidney disease. At this time, it is not known whether boosting mitochondria health and function in humans could reduce the harm of instability in blood pressure.

This research study is being done to try to explore the impact of HIRRT on mitochondria health and kidney recovery by assessing critically ill patients with AKI who are undergoing SLED treatment in ICU at The Ottawa Hospital.

DETAILED DESCRIPTION:
BACKGROUND:

Acute kidney injury (AKI) that requires renal replacement therapy (RRT) affects 2% of all hospitalized patients and 15% of those admitted to ICU. Non-recovery of kidney function and consequent long-term dialysis-dependence, has a profoundly negative impact on patients' health and quality of life.

While RRT is life-saving treatment for severe AKI, hemodynamic instability related to RRT (HIRRT) occurs frequently during all forms of RRT used in ICU. For slow low-efficiency dialysis (SLED), the RRT modality used for hemodynamically unstable patients at The Ottawa Hospital, HIRRT occurs during up to 86% of treatments. HIRRT may cause repetetive ischemia-reperfusion injury (IRI) to patients' already injured kidneys and may limit kidney recovery.

At the cellular level, after IRI, there is pronounced loss and dysfunction of mitochondria. Mitochondria are the organelles that serve as the primary source of energy to maintain cellular function. Their depletion and dysfunction results in the evolution of AKI to fibrosis and limits recovery of kidney function. The health of mitochondria depends greatly on a metabolite called nicotinamide adenine dinucleotide (NAD+). Animal studies and a recent phase 1 trial suggest that boosting NAD+ is a promising strategy to attenuate cardiac and kidney IRI. One potential NAD+ booster, nicotinamide riboside (NR), a NAD+ precursor, has an excellent safety profile after having undergone testing in multiple human trials for other indications.

Our group's recent systematic review found that few studies have assessed interventions to mitigate HIRRT in critically ill patients and that none targeted or assessed mitochondrial function. Whether boosting mitochondrial function is a truly a promising strategy for mitigating the harms of HIRRT depends on several unknowns. It remains to be determined if baseline levels of NAD+ and NAD+-related biomarkers (NRBs) in patients starting RRT are diminished and if these levels are affected by HIRRT.

Similarly, it is unknown if NAD+ and other NRB are removed from the blood by RRT itself.

OBJECTIVES:

Primary objective: Determine the levels of NAD+ and other NRBs before and after SLED treatments.

Secondary objectives: Determine if changes in NAD+ and other NRBs relate to the occurrence of HIRRT. Determine if SLED removes NAD+ and other NRBs by measuring dialysate levels.

EXPERIMENTAL PLAN: The investigators propose a prospective feasibility cohort study to measure and compare the levels of NAD+ and NRBs in AKI patients who are treated with SLED in ICU. The investigators conservatively estimate being able to recruit 60 patients over 2 years. Clinical data, as well as blood and urine samples will be obtained pre- and post-SLED for up to 3 consecutive treatments. Additional samples of dialysate will be tested to assess the extent to which NAD+ and NRBs are cleared by SLED.

SIGNIFICANCE: Elucidating the role of NAD+ or NRB in the kidney recovery of AKI patients who require RRT in ICU could lead to studies examining NAD+ boosting compounds' potential to mitigate HIRRT and improve clinical outcomes such as kidney recovery to RRT-independence. This approach has fewer barriers than there would be for developing a new NAD+-boosting compound as NR is already sold as a food supplement.

ELIGIBILITY:
Inclusion Criteria:

* >/=18 years;
* Diagnosis of stage 3 AKI per Kidney Disease Improving Global Outcomes (KDIGO) AKI guidelines;
* Starting SLED as first RRT received during current hospitalization.

Exclusion Criteria:

* Prior kidney transplant;
* Prior nephrectomy;
* Any RRT in the previous year;
* Baseline estimated glomerular filtration rate (eGFR) <15ml/min/1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AKI patients who are treated with SLED in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean arterial pressure (MAP) | 24 months
  Decline in MAP >=20 mmHg from the start of SLED or initiation of/increased dose of vasopressors required during SLED, occurring once or more during the SLED session.

SECONDARY OUTCOMES:
Frequency of HIRRT | 24 months
  Frequency of HIRRT according to primary outcome; death; kidney recovery to RRT-independence at time of hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada